CLINICAL TRIAL: NCT03296657
Title: A Pilot Study to Evaluate Stannous Fluoride in GCF and Subgingival Plaque
Brief Title: Analysis of Stannous Fluoride in GCF and Subgingival Plaque
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CSD2017123
Record Dates: First submitted 2017-09-13; First posted 2017-09-28 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Subgingival Plaque; GCF
MeSH Terms: interventions — Tin Fluorides

STUDY DESIGN:
Intervention Model Description: subject will brush twice a day for 2 weeks with stannous fluoride paste for at least 1 minute
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- stannous fluoride toothpaste (Experimental): 0.454% stannous fluoride will be used twice a day, brushing for at least 1 minute for 2 weeks
  Interventions: Drug: stannous fluoride

INTERVENTIONS:
Drug: stannous fluoride — subjects will brush with paste twice daily for 2 weeks

SUMMARY:
The amount of stannous fluoride in GCF and subgingival plaque samples will be analyzed.

DETAILED DESCRIPTION:
This is pilot study involving approximately 20 subjects with at least 20 dental pockets between 2- 4mm with bleeding for sampling. Subjects will have up to 10 sites identified as "sampling sites" that will have supragingival plaque, subgingival plaque, and gingival crevicular fluid (GCF) collected at Baseline, 30 minutes, 24 hours, and Week 2.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent to participate in the study;
* Be 18 years of age or older;
* Agree not to participate in any other oral/dental product studies during the course of this study;
* Agree to delay any elective dentistry (including dental prophylaxis) until the study has been completed;
* Agree to use the acclimation products and to refrain from using any other oral care products (including floss and mouth rinse) between the Acclimation and Baseline Visit;
* Agree to use the treatment products and refrain from any form of non-specified oral hygiene during the treatment periods (after the Baseline Visit), including but not limited to the use of products such as floss, mouth rinse, or whitening products;
* Agree to return for all scheduled visits and follow study procedures;
* Must have at least 16 natural teeth;
* Be in good general health, as determined by the Investigator/designee based on a review of the health history/update for participation in the study;
* Agree to refrain from all oral hygiene after 11 p.m. the night prior to each visit;
* Agree to refrain from eating, chewing gum, drinking and using tobacco for 4 hours prior to each visit;
* Have minimum 20 sampling sites with bleeding and pocket depth ≥2mm but not deeper than 4mm.

Exclusion Criteria:

* Having a dental prophylaxis within 2 weeks of Acclimation visit;
* Having rampant caries, open or untreated caries, or advanced periodontitis requiring prompt treatment;
* A medical condition requiring an antibiotic prophylaxis prior to dental visits;
* A history of hypersensitivity to oral care products containing stannous fluoride; or
* Have any condition or disease, as determined by the Investigator/Designee based on a review of the medical history, which could be expected to interfere with examination procedures or with the subject's safe completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-08-23 (Actual); Primary Completion 2017-09-22 (Actual); Study Completion 2017-09-22 (Actual)

PRIMARY OUTCOMES:
Amount of tin in GCF sample | mean difference from 30 minutes to baseline
  per GCF sample amount of stannous level in ng/uL will be measured

SECONDARY OUTCOMES:
Amount of tin in GCF and Subgingival Plaque | change from visit (change from 24 hours to baseline, change Week 2 to baseline)
  stannous level in subgingival plaque will be measured as concentration in ng, per GCF sample amount of stannous level in ng/uL

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Milleman, Principal Investigator — Salus Research
Locations (1):
- Salus Research, Fort Wayne, Indiana, United States